CLINICAL TRIAL: NCT01871402
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Comparison of 000-0551 Lotion Versus Vehicle Lotion in Subjects With Plaque Psoriasis (Study -304)
Brief Title: A Comparison of 000-0551 Lotion Versus Vehicle Lotion in Subjects With Plaque Psoriasis (Study -304)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000-0551-304
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis; lotion; investigator's global assessment
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Experimental): Topical lotion, applied twice daily
  Interventions: Drug: 000-0551 Lotion
- Vehicle Arm (Placebo Comparator): Topical lotion, applied twice daily
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: 000-0551 Lotion
  Arms: Active Arm
Drug: Vehicle Lotion
  Arms: Vehicle Arm

SUMMARY:
This Phase 3 study has been designed to determine and compare the efficacy and safety of 000-0551 Lotion and Vehicle Lotion applied twice daily for two weeks in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than 12% affected body surface area.
* Subject has an Investigator's Global Assessment (IGA) score of at least three (moderate) at study start.
* If subject is a woman of childbearing potential, she must have a negative urine pregnancy test and agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
* Subject has used any phototherapy (including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days prior to study start.
* Subject has used any systemic methotrexate, retinoids, systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids], cyclosporine or analogous products within 90 days prior to study start.
* Subject has used any systemic biologic therapy (i.e., FDA-approved or experimental therapy) within five half-lives of the biologic prior to study start.
* Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to study start or is intending to have such exposure during the study.
* Subject has used topical body (excluding the scalp) psoriasis therapy (including coal tar, anthralin, steroids, retinoids, vitamin D analogs) within 14 days prior to study start.
* Subject has used emollients/moisturizers on areas to be treated within four hours prior to clinical evaluation at study start.
* Subject is currently using lithium or Plaquenil (hydroxychloroquine).
* Subject is currently using a beta-blocking medication (e.g., propanolol) or angiotensin converting enzyme (ACE) inhibitor at a dose that has not been stabilized.
* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has used an investigational drug or investigational device treatment within 30 days prior to study start.
* Subject has been previously enrolled in this study and treated with a test article.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, Ph.D., Study Director — Therapeutics, Inc.
Locations (10):
- United States (10):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - UCSD Dermatology, San Diego, California
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Research Across America, Dallas, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 2013 to December 2013
  The location of clinical sites included dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Groups:
- Active Arm: Topical lotion, applied twice daily
  000-0551 Lotion
- Vehicle Arm: Topical lotion, applied twice daily
  Vehicle Lotion
Period: Overall Study
Arm/Group | Active Arm | Vehicle Arm
Started | 110 | 111
Completed | 109 | 108
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Vehicle Arm | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.28) | 50.8 (14.15) | 51.8 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 63 | 65 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 15 | 20
  Not Hispanic or Latino | 105 | 96 | 201
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 11 | 10 | 21
  White | 88 | 87 | 175
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 111 | 221

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Rated a "Treatment Success" Based on the Investigator's Global Assessment (IGA)
Description: The IGA score is a static evaluation of the overall or "average" degree of severity of a subject's disease, taking into account all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. IGA is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 15
Population: Analysis shown is based on the Intent-to-Treat population, defined as all enrolled participants who were randomized and applied at least one dose of the test article.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 110 | 111
percentage of participants | 44.5 | 6.3
Statistical Analysis 1: Comparison: Active Arm vs Vehicle Arm; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Treatment groups were compared with respect to the proportions of subjects with "treatment success" at Day 15 using the Cochran-Mantel-Haenszel (CMH) test stratified by analysis center; Multiple imputation was used to impute missing data from the ITT population

2. Secondary Outcome: Proportion of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: A static assessment of the overall or "average" degree of severity of each of three key characteristics present within all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. Each clinical sign of psoriasis is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 15
Population: Analysis shown is based on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 110 | 111
percentage of participants
  Scaling | 55.5 | 10.8
  Erythema | 36.4 | 7.2
  Plaque Elevation | 45.5 | 8.1
Statistical Analysis 1: Comparison: Active Arm vs Vehicle Arm; Treatment groups were compared with respect to each of the clinical signs of psoriasis (scaling, erythema, and plaque elevation); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance (<0.001) was achieved for each of the clinical signs of psoriasis (scaling, erythema, and plaque elevation); Missing data was imputed as treatment failure

3. Other Pre Specified Outcome: Proportion of Subjects With IGA "Treatment Success" at Day 8
Description: Interim analysis of IGA. "Treatment success" and IGA as defined in the primary outcome measure.
Time Frame: Day 8
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 109 | 110
percentage of participants | 16.5 | 1.8
Statistical Analysis 1: Comparison: Active Arm vs Vehicle Arm; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Other Pre Specified Outcome: Proportion of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis at Day 8
Description: Interim analysis of clinical signs of psoriasis (scaling, erythema and plaque elevation). "Treatment success" and clinical signs as defined in the secondary outcome measure.
Time Frame: Day 8
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 109 | 110
percentage of participants
  Scaling | 33.9 | 6.4
  Erythema | 13.8 | 0.9
  Plaque Elevation | 21.1 | 3.6
Statistical Analysis 1: Comparison: Active Arm vs Vehicle Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance (<0.001) was achieved for each of the clinical signs of psoriasis (scaling, erythema, and plaque elevations)

5. Other Pre Specified Outcome: Change From Baseline in Pruritus Score at Day 15
Description: Pruritus scale will be used to assess the subjective and multidimensional experience of the subject's pruritus (itching) during the previous two weeks at Baseline and Day 15. Possible scores range from 5 (no pruritus) to 25 (most severe pruritus).
Time Frame: Baseline and Day 15
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 109 | 107
units on a scale | -5.2 (3.46) | -3.1 (3.35)

6. Other Pre Specified Outcome: Change in % Body Surface Area (BSA) With Active Psoriasis at Days 8 and 15
Description: The investigator will use the assumption that 1% BSA is approximately equal to the surface area of the subject's palm and fingers, with the fingers extended yet grouped together, creating a flat oval-like surface area.
Time Frame: Baseline, Day 8 and Day 15
Population: Analysis shown is based on the ITT population at Days 8 and 15 and compared to baseline. Number of Participants Analyzed is at Day 15; at Day 8, N=109 (Active) and N=110 (Vehicle). Only participants with observed values are reported.
Measure: Mean (Standard Deviation); unit: Change in %BSA
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 109 | 108
Change in %BSA
  Day 8 | -0.7 (1.59) | -0.1 (0.73)
  Day 15 | -1.6 (2.22) | -0.2 (1.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 15) or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The Safety population included all subjects enrolled in the study who were dispensed the test article at least once; because the first dose of the test article was applied at the study site (Day 1), all enrolled subjects (N=221) were included in the safety population. Most AEs were mild in severity.
Arm/Group | Active Arm | Vehicle Arm
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/111
Other Adverse Events (participants affected / at risk) | 2/110 | 7/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=110) | Vehicle Arm (N=111)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 0 (0) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.